CLINICAL TRIAL: NCT07219368
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Doses of MT-201 in Healthy Participants
Brief Title: A First-in-Human Single and Multiple Ascending Dose Study of MT-201
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mirador Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: MT-201-101
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer
Keywords: MT-201; Phase 1
MeSH Terms: interventions — adecatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose of MT-201 (Experimental): To assess the safety and tolerability of single intravenous/subcutaneous doses of MT-201
  Interventions: Drug: MT-201
- Multiple Ascending Dose of MT-201 (Experimental): To assess the safety and tolerability of multiple intravenous/subcutaneous doses of MT-201
  Interventions: Drug: MT-201
- Single Ascending Dose Placebo Arm (Placebo Comparator): To assess the safety and tolerability of single intravenous/subcutaneous doses of placebo
  Interventions: Drug: Placebo
- Multiple Ascending Dose Placebo (Placebo Comparator): To assess the safety and tolerability of multiple intravenous/subcutaneous doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-201 — MT-201
  Arms: Multiple Ascending Dose of MT-201; Single Ascending Dose of MT-201
Drug: Placebo — Placebo
  Arms: Multiple Ascending Dose Placebo; Single Ascending Dose Placebo Arm

SUMMARY:
First-in-human study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single and multiple doses of MT-201 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male participant or female participant of nonchildbearing potential between 19 and 55 years of age (inclusive) at the time of signing informed consent.
2. Female participants must be of nonchildbearing potential, defined as postmenopausal or surgically sterile, and have official documentation, at least 6 months prior to the first dose.
3. Male participants with female partners of childbearing potential who are involved in heterosexual intercourse or activities that could lead to pregnancy must use barrier method of contraception (male condom) and refrain from sperm donation.
4. Good general health.
5. Able to provide written informed consent and understand and comply with the requirements of the study.

Exclusion Criteria:

1. History or presence of any clinically significant organ system disease.
2. Abnormal laboratory assessments, physical exam of ECG outside the normal range that is judged by the Investigator to be clinically significant.
3. History of alcohol or drug abuse within the past 24 months.
4. Current use or history of regular tobacco, or nicotine-containing products within 3 months prior to screening.
5. Administration or use of any investigational drug or device within 30 days preceding the first dose of study drug administration.
6. Blood donation within 60 days prior to dosing or plasma donation within 14 days prior to dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male and female (of non-childbearing potential only)
Enrollment: 72 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with non-SAEs and SAES | Up to 40 weeks
  Incidence of adverse events, clinically significant laboratory abnormalities, clinically significant electrocardiogram, vital signs, and physical examination abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirador Clinical Department, San Diego, California 92121, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No